CLINICAL TRIAL: NCT06017427
Title: Evaluation of Patient Satisfaction During Treatment With Dupilumab in Severe and Recurrent Nasosinusal Polyposis Despite Appropriate Medical and Surgical Treatment.
Acronym: Dupi-PNS
Status: Terminated | Type: Observational
Why Stopped: Number of inclusions sufficient for answering the main objective
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Other Study IDs: 22-005
Record Dates: First submitted 2023-07-18; First posted 2023-08-30 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
Keywords: CRSwNP; decreased quality of life; Nasal polyps; Rhinosinusitis; recurrent CRSwNP; severe CRSwNP
MeSH Terms: conditions — Nasal Polyps; Rhinosinusitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suffering from severe recurrent CRSwNP and treated with Dupilumab: Patients suffering from severe recurrent CRSwNP despite having benefited from the appropriate medical and surgical treatment and treated with Dupilumab for 6 months
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Submission of several questionnaires (Quality of Life and clinical scores) at three time points: before initiation of Dupilumab, after 6 months of Dupilumab treatment, and 6 months after stopping Dupilumab treatment

SUMMARY:
Chronic rhinosinusitis with nasal polyps (CRSwNP) or nasal polyposis is a frequent disease leading to a decreased quality of life. The validated course of treatment is firstly a medical one with saline irrigations and topical corticosteroids, followed by surgery (ethmoidectomy) if the medical treatment fails.

In many cases, CRSwNP becomes a recurrent disease despite maximal treatment as previously indicated and it becomes refractory, with a chronically reduced quality of life.

New treatments known as Biologics or Biotherapies in France such as Dupilumab are now available in situations of severe recurrent CRSwNP despite the appropriate treatment.

The goal of this study is to assess the clinical effectiveness of Dupilumab and patient satisfaction, in a cohort of french patients, focusing on the change in quality of life that is expected from said treatment, over a period of one year.

Patients will undergo 6 months of treatment with Dupilumab, the treatment will then be stopped for the next 6 months.

The primary judgment criteria will be the SNOT 22 score, measured before treatment, after 6 months of treatment, and 6 months after stopping treatment, over a telephonic conversation.

DETAILED DESCRIPTION:
CRSwNP has existed for over 5000 years, it is a frequent disease, affecting 1 to 4 % of the general population, especially older men and is defined by inflammatory modification of the sinuses and nasal cavities with benign growths of the mucosa known as polyps. It leads to numerous symptoms (nasal blockage, anosmia, nasal dripping, fatigue, pain), which have important consequences in terms of quality of life, social interactions, and by the heavy costs that are brought by medical and surgical treatment.

It is a multifactorial disease for which physiopathology is not well established.

No definitive treatment exists. The appropriate course of treatment aims to control the disease, but not cure it, via topical corticosteroids application which can be facilitated by endoscopic surgery (polypectomy, ethmoidectomy).

Recurrence is frequent after surgery (40 %, 18 months after surgery), which leads to more surgeries that get more complicated and riskier each time.

CRSwNP is also an expensive disease (several thousands of euros per year for one patient), especially in cases of recurrence after surgical treatment. The indirect costs are also high with work absenteeism and decreased productivity making CRSwNP one of the 10 most costly diseases for US employers.

Dupilumab, a biologic treatment targeting the receptors of IL4 and IL13 which are major actors of the inflammatory reaction at hand in CRSwNP, has recently appeared on the market for treatment of severe recurrent CRSwNP despite the appropriate medical and surgical treatment, and has proved its efficacy in randomized clinical trials.

It is a very expensive treatment (1400 euros a month for one patient in France), which is why its clinical effectiveness in a real-life setting must be assessed.

Hypothesis : Dupilumab improves symptoms and quality of life in severe recurrent CRSwNP despite the appropriate medical and surgical treatment.

Objectives : To assess the effect of Dupilumab and patient satisfaction during treatment and after its discontinuation, on symptoms and quality of life in patients suffering from severe and recurrent CRSwNP despite having benefited from the appropriate medical and surgical treatment, in a French real-life cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men over 18 years old
2. Suffering from severe and recurrent Chronic Rhinosinusitis with Nasal Polyps despite having benefited from the appropriate medical and surgical treatment.
3. CRSwNP diagnosis established on the basis of clinical presentation and patient interrogation by their referent ENT surgeon.
4. Patient treated with Dupilumab in the indication depicted in bullet point 2.
5. Patient having voiced their non-opposition to this research, having received clear and appropriate information.
6. Patient affiliated to the French Social Security.

Exclusion Criteria:

1. Patient having undergone endoscopic nasal surgery during their Dupilumab treatment.
2. Patient presenting exclusion criteria for Dupilumab treatment.
3. Patient suffering from immune deficit.
4. Patient suffering from vascularitis with nasal expression.
5. Patient whose autonomy has been reduced by a legal authority.
6. Patient unable to express their agreement to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, men or women, of any age, having received treatment with Dupilumab for the indication of recurrent severe nasal polyposis despite surgery and appropriate medical treatment
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Assessment of the global effect of Dupilumab 1 day before Dupilumab by the mean of the SNOT 22 score | 1 day before Dupilumab
  The SNOT22 score is a validated questionnaire for the assessment of symptoms of Chronic rhinosinusitis, ranging from 0 to 110. The more severe are the disease and its associated symptoms, the higher is the score
Assessment of the global effect of Dupilumab 6 months of Dupilumab treatment by the mean of the SNOT 22 score | 6 months of Dupilumab treatment
  The SNOT22 score is a validated questionnaire for the assessment of symptoms of Chronic rhinosinusitis, ranging from 0 to 110. The more severe are the disease and its associated symptoms, the higher is the score
Assessment of the global effect of Dupilumab 6 months after stopping the treatment by the mean of the SNOT 22 score | 6 months after stopping Dupilumab treatment
  The SNOT22 score is a validated questionnaire for the assessment of symptoms of Chronic rhinosinusitis, ranging from 0 to 110. The more severe are the disease and its associated symptoms, the higher is the score

SECONDARY OUTCOMES:
Assessment of the effect of Dupilumab on nasal obstruction by the mean of the Visual Analogic Scale for nasal obstruction | 1 day before Dupilumab, at 6 months of Dupilumab treatment, and 6 months after stopping Dupilumab treatment
  Staging nasal obstruction level from 0 to 10. The more severe are the symptoms, the higher is the score
Assessment of the effect of Dupilumab on the olfaction by the mean of the Visual Analogic Scale for Olfaction | 1 day before Dupilumab, at 6 months of Dupilumab treatment, and 6 months after stopping Dupilumab treatment
  Staging olfaction levels from 0 to 10. The more severe are the symptoms, the higher is the score
Assessment of the effect of Dupilumab on the severity of the nasal polyposis by the mean of the Nasal Polyp Score | 1 day before Dupilumab, at 6 months of Dupilumab treatment, and 6 months after stopping Dupilumab treatment
  Endoscopic based score assessing the severity of nasal polyposis, 0 to 8. The more severe are the symptoms, the higher is the score
Assessment of the effect of Dupilumab on the severity of the nasal polyposis on an iconographic level by the mean of the Lund McKay score | 1 day before the treatment initiation
  CT-scan based score assessing the severity of nasal polyposis on an iconographic level, 0 to 24. The more severe are the symptoms, the higher is the score
Assessment of the effect of Dupilumab on the quality of life by the mean of the EQ 5D 5L score | 1 day before Dupilumab, at 6 months of Dupilumab treatment, and 6 months after stopping Dupilumab treatment
  Quality of life questionnaire associated with a Visual Analogic Scale ranging from 0 to 100. The more severe are the symptoms, the higher is the score
Assessment of the effect of Dupilumab on the severity of the asthma by the mean of the ACT score | 1 day before Dupilumab, at 6 months of Dupilumab treatment, and 6 months after stopping Dupilumab treatment
  Asthma control assessment score ranging from 5 to 25. The more severe are the symptoms, the higher is the score
Assessment of the time to first improvement in sense of smell and nasal obstruction with Dupilumab | 1 day
  Time between the beginning of treatment with Dupilumab and the first time a reduction in nasal obstruction and hyposmia was observed by the patient
Time between stopping Dupilumab and possible deterioration of the sense of smell and nasal obstruction | 1 day
  Time between the stopping of Dupilumab treatment and the first worsening of nasal obstruction and olfaction that was noted by the patient
Evolution of a potential middle ear chronic inflammation during treatment | 1 day
  rate of otitis appearance among the patients during their treatment with Dupilumab
Necessity to use oral corticosteroids during or after Dupilumab treatment | 1 day
  Rate of patients in need of corticosteroids during or after their treatment with Dupilumab
Evolution to nasosinus superinfections during and after Dupilumab treatment | 1 day
  Rate of nasosinus superinfections appearance observed during or after the treatment with Dupilumab
Collect of adverse effects during Dupilumab treatment | 1 day
  collect of adverse effects during Dupilumab treatment

CONTACTS AND LOCATIONS:
Overall Officials: Léa FATH, MD, PhD, Principal Investigator — HUS
Locations (1):
- Hautepierre Hospital, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Settipane RA, Peters AT, Chiu AG. Chapter 6: Nasal polyps. Am J Rhinol Allergy. 2013 May-Jun;27 Suppl 1:S20-5. doi: 10.2500/ajra.2013.27.3926. PMID 23711034
- [Background] Stjarne P, Odeback P, Stallberg B, Lundberg J, Olsson P. High costs and burden of illness in acute rhinosinusitis: real-life treatment patterns and outcomes in Swedish primary care. Prim Care Respir J. 2012 Jun;21(2):174-9; quiz 10p following 179. doi: 10.4104/pcrj.2012.00011. PMID 22349918
- [Background] Teul I, Zbislawski W, Baran S, Czerwinski F, Lorkowski J. Quality of life of patients with diseases of sinuses. J Physiol Pharmacol. 2007 Nov;58 Suppl 5(Pt 2):691-7. PMID 18204184
- [Background] Hopkins C, Browne JP, Slack R, Lund V, Topham J, Reeves B, Copley L, Brown P, van der Meulen J. The national comparative audit of surgery for nasal polyposis and chronic rhinosinusitis. Clin Otolaryngol. 2006 Oct;31(5):390-8. doi: 10.1111/j.1749-4486.2006.01275.x. PMID 17014448
- [Background] Leopold DA, Elkayam D, Messina JC, Kosik-Gonzalez C, Djupesland PG, Mahmoud RA. NAVIGATE II: Randomized, double-blind trial of the exhalation delivery system with fluticasone for nasal polyposis. J Allergy Clin Immunol. 2019 Jan;143(1):126-134.e5. doi: 10.1016/j.jaci.2018.06.010. Epub 2018 Jun 19. PMID 29928924
- [Background] Kobayashi Y, Yasuba H, Asako M, Yamamoto T, Takano H, Tomoda K, Kanda A, Iwai H. HFA-BDP Metered-Dose Inhaler Exhaled Through the Nose Improves Eosinophilic Chronic Rhinosinusitis With Bronchial Asthma: A Blinded, Placebo-Controlled Study. Front Immunol. 2018 Sep 25;9:2192. doi: 10.3389/fimmu.2018.02192. eCollection 2018. PMID 30337921
- [Background] Rice DH. Endoscopic sinus surgery. Otolaryngol Head Neck Surg. 1994 Jul;111(1):100-10. doi: 10.1177/019459989411100118. No abstract available. PMID 8028915
- [Background] Benninger MS, Sindwani R, Holy CE, Hopkins C. Impact of medically recalcitrant chronic rhinosinusitis on incidence of asthma. Int Forum Allergy Rhinol. 2016 Feb;6(2):124-9. doi: 10.1002/alr.21652. Epub 2015 Dec 1. PMID 26624856
- [Background] DeConde AS, Mace JC, Levy JM, Rudmik L, Alt JA, Smith TL. Prevalence of polyp recurrence after endoscopic sinus surgery for chronic rhinosinusitis with nasal polyposis. Laryngoscope. 2017 Mar;127(3):550-555. doi: 10.1002/lary.26391. Epub 2016 Nov 12. PMID 27859303
- [Background] Bhattacharyya N. Contemporary assessment of the disease burden of sinusitis. Am J Rhinol Allergy. 2009 Jul-Aug;23(4):392-5. doi: 10.2500/ajra.2009.23.3355. PMID 19671253
- [Background] Wahid NW, Smith R, Clark A, Salam M, Philpott CM. The socioeconomic cost of chronic rhinosinusitis study. Rhinology. 2020 Apr 1;58(2):112-125. doi: 10.4193/Rhin19.424. PMID 32172284
- [Background] Lourijsen ES, Fokkens WJ, Reitsma S. Direct and indirect costs of adult patients with chronic rhinosinusitis with nasal polyps. Rhinology. 2020 Jun 1;58(3):213-217. doi: 10.4193/Rhin19.468. PMID 32415826
- [Background] Bhattacharyya N. Assessing the additional disease burden of polyps in chronic rhinosinusitis. Ann Otol Rhinol Laryngol. 2009 Mar;118(3):185-9. doi: 10.1177/000348940911800305. PMID 19374149
- [Background] Goetzel RZ, Hawkins K, Ozminkowski RJ, Wang S. The health and productivity cost burden of the "top 10" physical and mental health conditions affecting six large U.S. employers in 1999. J Occup Environ Med. 2003 Jan;45(1):5-14. doi: 10.1097/00043764-200301000-00007. PMID 12553174
- [Background] Rudmik L. Economics of Chronic Rhinosinusitis. Curr Allergy Asthma Rep. 2017 Apr;17(4):20. doi: 10.1007/s11882-017-0690-5. PMID 28337570
- [Background] Bachert C, Mannent L, Naclerio RM, Mullol J, Ferguson BJ, Gevaert P, Hellings P, Jiao L, Wang L, Evans RR, Pirozzi G, Graham NM, Swanson B, Hamilton JD, Radin A, Gandhi NA, Stahl N, Yancopoulos GD, Sutherland ER. Effect of Subcutaneous Dupilumab on Nasal Polyp Burden in Patients With Chronic Sinusitis and Nasal Polyposis: A Randomized Clinical Trial. JAMA. 2016 Feb 2;315(5):469-79. doi: 10.1001/jama.2015.19330. PMID 26836729